CLINICAL TRIAL: NCT01235312
Title: Microcirculatory Mapping of the Aging Hand and Foot
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Hannover Medical School, Plastic, Hand and Reconstructive Surgery, Hannover Medical School, Plastic, Hand and Reconstructive Surgery
Other Study IDs: Kraemer003
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Cutaneous Microcirculation in Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Healthy subjects
- Patients suffering from Diabetes mellitus
- Patients suffering from peripheral arterial occlusive disease

SUMMARY:
Currently, dorsal hand rejuvenation is an upcoming issue as patients seek plastic surgeons to address this highly visible area, although no specific statistics concerning the number of patients undergoing dorsal hand rejuvenation have been published yet. The solitary use of fillers, fat, sclerotherapy, skin excision, resurfacing and combinations of the above mentioned therapies have been reported in the literature, but still there is a lack of scientific literature about functional microcirculation of the dorsum of the hand.

Furthermore, there is a lack of scientific data about functional microcirculation of the plantar foot in healthy subjects compared to patients suffering from Diabetes mellitus or peripheral arterial occlusive disease. Consequently, the aim of this study is the evaluation of the functional microcirculation of hands and feet in healthy subjects as well as patients suffering from the above mentioned diseases.

ELIGIBILITY:
Inclusion Criteria:

* Both healthy subjects and patients suffering from diabetes mellitus or manifested peripheral arterial occlusive disease aged between 18 and 75 years

Exclusion Criteria:

* soft tissue inflammation or osteomyelitis, liver disease, cardiac dysfunction, arterial hypotension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both healthy subjects and patients suffering from diabetes mellitus or manifested peripheral arterial occlusive disease
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Correlation of microcirculation to age and incidence of vascular diseases | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Hannover, Hanover, Germany